CLINICAL TRIAL: NCT00487461
Title: Randomized Double Blind Study Using Simvastatin for the PRevention Aof Vasospasm in Aneurysmal Subarachnoid Hemorrhage
Brief Title: Use of Simvastatin for the Prevention of Vasospasm in Aneurysmal Subarachnoid Hemorrhage
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study PI left the institution and study was stopped at that time.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ali Alaraj, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2005-0857
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Cerebral Vasospasm
Keywords: SAH; Vasospasm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — Simvastatin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo
- Study Group #1 (Experimental): Simvastatin 40 mg
  Interventions: Drug: Simvastatin 40 mg
- Study Group #2 (Experimental): Simvastatin 80 mg
  Interventions: Drug: Simvastatin 80 mg

INTERVENTIONS:
Drug: Simvastatin 40 mg — Comparing two doses of Simvastatin to placebo
  Other Names: Zocor
  Arms: Study Group #1
Drug: Placebo — Placebo tablet
  Other Names: dummy pill, sugar pill
  Arms: Control Group
Drug: Simvastatin 80 mg — Comparing two doses of Simvastatin to placebo
  Other Names: Zocor
  Arms: Study Group #2

SUMMARY:
The purpose of this study is to test whether treatment with a drug called Simvastatin prevents and improves outcome in patients who have Subarachnoid bleeding. Simvastatin is currently approved for the treatment of high cholesterol levels.

DETAILED DESCRIPTION:
Aneurysmal Subarachnoid hemorrhage or SAH (bleeding on the surface of the brain) affects 10 per 100,000 population each year. For survivors of the initial hemorrhage, delayed narrowing of the blood vessels (vasospasm) and related delayed strokes are the most common serious complication. Narrowing of blood vessels affect 30% of patients with such bleeding. Despite maximum therapy, nearly 50% of patients with symptomatic vasospasm with develop stroke. Because cerebral vasospasm remains the leading cause of morbidity and mortality after aSAH, this critically important issue needs further studies.

One hundred and fifty patients will be randomized, 50 to each arm of the study. Patients enrolled in the study will be receive the drug (either Simvastatin 40 mg or Simvastatin 80 mg per mouth daily), while the control group will receive a sugar tablet. The treatment will be continued for a total of 21 days. The neurological abilities (Stroke Outcome measures, these are included with the application for your review) at day 21 post aSAH will be reviewed at time of discharge as well at 6 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old inclusive
* Subarachnoid hemorrhage diagnosed by CT on admission
* Randomizable within 732 hours of subarachnoid hemorrhage
* Saccular intracranial aneurysm proven by cerebral angiography or computed tomographic angiography (CTA)
* Surgical or endovascular obliteration
* Able to obtain written informed consent from patient or surrogate

Exclusion Criteria:

* Pregnancy, as confirmed by routine urine test on admission
* Elevated liver function test at time of randomization, defined as more than three times the upper limit of normal
* On Statins, niacin, or fibrate therapy within 30 days of presentation
* Any vasospasm on the initial diagnostic angiogram
* Glasgow Coma Scale 5 or less at the time of randomization
* History of liver disease or active liver disease
* Hypersensitivity to statins
* Patient taking medication not recommended for concomitant use with Simvastatin (40 or 80 mg) as per the product label

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Z. Roitberg, MD, Principal Investigator — Assnt Prof. Univ. of Illinois at Chicago, Dept of Neurosurgery; Ali Alaraj, MD, Principal Investigator — Clinical Fellow Department of Neurosurgery
Locations (1):
- Univeristy of Illinois at Chicago, Dept of Neurosurgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group #1: Simvastatin 40 mg
  Simvastatin: Comparing two doses of Simvastatin to placebo
- Study Group #2: Simvastatin 80 mg
  Simvastatin: Comparing two doses of Simvastatin to placebo
Period: Overall Study
Arm/Group | Control Group | Study Group #1 | Study Group #2
Started | 2 | 12 | 11
Completed | 2 | 10 | 7
Not Completed | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group #1 | Study Group #2 | Total
Number analyzed (Participants) | 2 | 12 | 11 | 25
Age, Continuous [Median (Standard Deviation); unit: years] | 57 (5.6) | 47 (10.7) | 50 (11.6) | 49 (10.9)
Age, Customized [Number; unit: participants]
  > 70 years | 0 | 1 | 2 | 3
  60-70 years | 1 | 0 | 1 | 2
  50-60 years | 1 | 3 | 3 | 7
  40-50 years | 0 | 6 | 4 | 10
  < 40 years | 0 | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 8 | 18
  Male | 0 | 4 | 3 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 1 | 6 | 4 | 11
  Black | 0 | 3 | 4 | 7
  Hispanic | 1 | 3 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 2 | 12 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: To Measure Outcome in Patients Diagnosed With Aneurysmal Subarachnoid Hemorrhage (aSAH) Treated With Simvastatin, by Assessing Neurological Outcome by Accessing Glasgow Outcome Score, Modified Rankin Scale, and Barthel Index Score at Day 21 Post aSAH
Time Frame: 21 days
Population: Study PI left before outcome data was collected for the study and therefore the Outcome(s) will never be analyzed.
Arm/Group | Control Group | Study Group #1 | Study Group #2
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: To Determine Efficiency of Simvastatin in Decreasing the Incidence of Clinical Vasospasm in aSAH, and Define the Optimal Dose of Simvastatin and to Measure Outcome at 6 Months Follow up
Description: Study PI left before the efficacy of Simvastatin decreasing the incidence of clinical vasospasm in aSAH, and defining the optimal dose of Simvastatin and measuring the outcome at 6 months follow up data was collected for the study and therefore these outcomes will never be analyzed.
Time Frame: 6 months
Population: Study PI left before the efficacy of Simvastatin decreasing the incidence of clinical vasospasm in aSAH, and defining the optimal dose of Simvastatin and measuring the outcome at 6 months follow up data was collected for the study and therefore these outcomes will never be analyzed.
Arm/Group | Control Group | Study Group #1 | Study Group #2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed.
Arm/Group | Control Group | Study Group #1 | Study Group #2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed and Primary Physician leaving institution before study completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No